CLINICAL TRIAL: NCT03816709
Title: Intramuscular Heating Rates of a Chattanooga Intelect XT Therapeutic Ultrasound With 3 MHz, 1.0 W/cm2 at Three Depths up to 2.5 cm
Brief Title: Intramuscular Heating Rates of a Chattanooga Intelect XT Therapeutic Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Principal Investigator, Kara Gange, Associate Professor, North Dakota State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HE19132
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Ultrasound Therapy; Complications
Keywords: heating rates; therapeutic ultrasound
MeSH Terms: interventions — Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Therapeutic ultrasound treatment (Other): All subjects received a therapeutic ultrasound treatment with the Chattanooga Intelect Legend XT machine with the following parameters: 3 MHz, 1.0 W/cm2, 15 minute treatment time.
  Interventions: Device: Therapeutic Ultrasound

INTERVENTIONS:
Device: Therapeutic Ultrasound — A therapeutic ultrasound treatment was applied to the left medial gastrocnemius muscle with the following parameters: 3 MHz, 1.0 W/cm2 for 15 minutes.
  Other Names: Ultrasound therapy

SUMMARY:
The purpose of this study is to determine the rate of tissue temperature increase in the triceps surae during an ultrasound treatment using the Chattanooga Intelect Legend XT. The following parameters will be used: 3 MHz frequency, 1.0 W/cm2 intensity, 15 minute treatment time. Thermocouples will be inserted at 1.0, 1.75, and 2.5 cm depths to determine the heating rates. Most modality textbook recommendations for therapeutic ultrasound are based on studies performed with the Omnisound ultrasound machine. Previous research has shown variations in power output across manufacturers, producing differences in tissue temperature increases. No information has been published regarding the heating rates of the Chattanooga Intelect Legend XT machine for ultrasound treatments. By determining the heating rates for this machine, clinicians will be better able to utilize the Chattanooga Intelect Legend XT to help reach therapeutic goals.

DETAILED DESCRIPTION:
Individual subjects will report to the research lab. They will be instructed to wear appropriate shorts or pants that can be rolled up to expose the gastrocnemius (calf) muscle. The subject will lay prone on the treatment table with the foot and lower leg off of the treatment table in a relaxed, comfortable position. The following procedures will be completed using universal precautions:

1. The investigator will prep the treatment area by having the subject flex the calf to determine the proper location for the ultrasound treatment in the middle of the medial gastrocnemius muscle belly at its largest girth.

   1. A carpenter's square with markings along the vertical arm at the three experimental depths (1.0, 1.75, 2.5 cm) will be used.
   2. The horizontal arm of the carpenter's square will be covered in tape. The carpenter's square is then placed just proximal to the treatment mark while the level on the horizontal arm is used to maintain a level measure.
   3. Marks will be made on the muscle belly parallel to the marks on the vertical axis at 1.0, 1.75 and 2.5 cm depths.
   4. A mark is also made on the horizontal arm tape in line with the treatment mark on the medial gastrocnemius.
2. The Terason uSmart 3300 diagnostic ultrasound unit will be used to measure the adipose thickness over the treatment area and look for abnormalities in the treatment and thermocouple insertion areas. Aquasonic® 100 ultrasound gel will be placed on the 15L4 transducer. The transducer with gel will be placed over the mark of the treatment area. Once the transducer is in place, the screen will be frozen and the skin and adipose thickness will be measured using the caliper tool.
3. The thermocouples will be removed from the MetriCide after sterilizing for a minimum of 12 hours prior to insertion.

   1. The distal aspect of the thermocouple will be wiped dry with sterile gauze.
   2. A mark with a sharpie will be made on each thermocouple just past the length marked on the horizontal arm of the carpenter's square. This allows the tip of each thermocouple to be directly below the treatment site. A second mark will be made at 5 cm to make sure the thermocouple does not go too deep into the tissue.
   3. The distal end of the thermocouple will be wiped clean again using a 70% isopropyl alcohol wipe up to the marks and then the thermocouple will be wrapped in sterile gauze until it is inserted.
4. The insertion areas will be shaved to remove any body hair (if necessary) and cleaned using Betadine.

   a. Once the Betadine dries, 70% isopropyl alcohol will be wiped over the insertion area and given time to dry.
5. The subject will be instructed to take two deep breaths, while the researcher lightly grasps the gastrocnemius to confirm muscle relaxation.

   1. During the second exhalation, the 1.16 in needle catheter will be placed into the subject's calf at the 1.0 cm depth insertion mark using the level to guide the needle in. The needle will be removed leaving the catheter in the tissue.
   2. The thermocouple will be threaded through the catheter to the appropriate depth marked on the thermocouple and the catheter will be removed.
   3. The thermocouple will be secured using medical tape to keep it from moving.
   4. This procedure will be performed 3 times, with one thermocouple placed at each respective depth: 1.0 cm, 1.75 cm, and 2.5 cm.
6. Each thermocouple will be attached to the Iso Thermex electronic thermometer (Columbus Instruments, Columbus, OH), which will measure and record intramuscular temperatures from the tips of the thermocouples.
7. An ultrasound treatment template will be applied at the treatment site and secured with tape to maintain consistent treatment size.

   a. This template will be twice the size of the transducer's Effective Radiating Area (ERA).
8. A metronome will be utilized to consistently move the transducer at a rate of 4 cm/s .
9. The ultrasound treatment will begin once the intramuscular temperature has remained the same for a minute.
10. Each subject will receive one ultrasound treatment at the following parameters: 3 MHz frequency, 1.0 W/cm2 intensity, and 100% duty cycle using the Chattanooga Intelect® Legend XT.

    a. Termination of treatment will result when any of the following occur: i. A 15-minute treatment time is obtained. ii. A 4°C temperature increase occurs at all three depths as this has been shown as the necessary temperature change to increase tissue extensibility.

    iii. A 45°C temperature is reached at any depth, due to concern of tissue damage at high temperatures.

    iv. The subject experiences any pain or discomfort during the treatment.
11. Following the treatment, the ultrasound gel will be wiped from the leg, the template and thermocouples will be removed, and the insertion sites will be cleaned with 70% isopropyl alcohol wipes and covered with a band aid.
12. The subject will then be instructed on the possibility of minor soreness for the next day or two and instructed on an icing schedule to decrease discomfort.

ELIGIBILITY:
Inclusion Criteria:

* males and females between the ages of 18 - 35 years old
* able to speak English
* have less than 1 cm of adipose over the left medial gastrocnemius muscle.

Exclusion Criteria:

* any current lower extremity injury
* any lower extremity injuries within the last 6 months
* open wounds
* skin infections
* impaired circulation
* peripheral vascular disease
* deep vein thrombosis
* advanced arthritis
* poor thermal regulation
* anesthetic areas
* neoplasms/tumors
* thrombophlebitis
* closed infections
* any allergies or sensitivities to betadine
* any abnormalities observed in the medial gastrocnemius muscle determined by diagnostic ultrasound
* 1.0 cm or greater adipose over the left medial gastrocnemius muscle.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristy Shirley, Study Director — NDSU IRB
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No
Once the data has been analyzed to determine the heating rates, a manuscript including the heating rates will be submitted for publication.

REFERENCES:
- [Background] Gange KN, Kjellerson MC, Berdan CJ. The Dynatron Solaris(R) Ultrasound Machine: Slower Heating Than Textbook Recommendations at 3 MHz, 1.0 W/cm2. J Sport Rehabil. 2018 Jan 1;27(1):22-29. doi: 10.1123/jsr.2016-0173. Epub 2018 Jan 18. PMID 27992304
- [Background] Merrick MA, Bernard KD, Devor ST, Williams MJ. Identical 3-MHz ultrasound treatments with different devices produce different intramuscular temperatures. J Orthop Sports Phys Ther. 2003 Jul;33(7):379-85. doi: 10.2519/jospt.2003.33.7.379. PMID 12918863
- [Background] Draper DO, Castel JC, Castel D. Rate of temperature increase in human muscle during 1 MHz and 3 MHz continuous ultrasound. J Orthop Sports Phys Ther. 1995 Oct;22(4):142-50. doi: 10.2519/jospt.1995.22.4.142. PMID 8535471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-five subjects were recruited through the Institution's Listserve from January-February, 2019.
Period: Overall Study
Arm/Group | Therapeutic Ultrasound Treatment
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: male and female 18-35 year olds with no injuries to the lower leg.
Arm/Group | Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — 18-35 year olds
  Participants
    <=18 years | 0
    Between 18 and 65 years | 25
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Heating Rate at 1 cm Depth
Description: A thermocouple was inserted at the 1 cm depth to determine the tissue temperatures.
Time Frame: Baseline to end of treatment (up to 15 minutes or until temperatures increased 4 degrees, which occurred at 6 minutes)
Population: Intent to treat population. All subjects received the Ultrasound treatment with a thermocouple recording tissue temperatures at the 1 cm depth.
Measure: Mean (Standard Deviation); unit: degrees Celcius
Groups:
- Therapeutic Ultrasound Treatment: All subjects received a therapeutic ultrasound treatment with the Chattanooga Intelect Legend XT machine with the following parameters: 3 MHz, 1.0 W/cm2, 15 minute treatment time.
  Therapeutic Ultrasound: A therapeutic ultrasound treatment was applied to the left medial gastrocnemius muscle with the following parameters: 3 MHz, 1.0 W/cm2 for 15 minutes at the depths of 1.0, 1.75, and 2.5 cm.
Arm/Group | Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 25
degrees Celcius | 6.49 (1.24)

2. Primary Outcome: Heating Rate at 1.75 cm Depth
Description: A thermocouple was inserted at the 1.75 cm depth to determine the tissue temperatures.
Time Frame: Baseline to end of treatment (up to 15 minutes or until temperatures increased 4 degrees, which occurred at 8 minutes)
Population: Intent to treat. All subject received the Ultrasound treatment with a thermocouple at the 1.75 cm depth to determine tissue temperature
Measure: Mean (Standard Deviation); unit: degrees Celcius
Arm/Group | Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 25
degrees Celcius | 5.50 (1.34)

3. Primary Outcome: Heating Rate at 2.5 cm Depth
Description: A thermocouple was inserted at the 2.5 cm depth to determine the tissue temperatures.
Time Frame: Baseline to end of treatment (up to 15 minutes or until temperatures increased 4 degrees, which did not occur in the 15 minute treatment)
Population: Intent to treat. All subjects received the Ultrasound treatment with a thermocouple at the 2.5 cm depth to determine tissue temperatures.
Measure: Mean (Standard Deviation); unit: degrees Celcius
Arm/Group | Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 25
degrees Celcius | 3.07 (1.53)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Therapeutic Ultrasound Treatment
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03816709/Prot_005.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03816709/SAP_006.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03816709/ICF_007.pdf